CLINICAL TRIAL: NCT06623253
Title: Survey on Predictors of Discharge from Stroke Units in Argentina
Brief Title: Survey Stroke Units in Argentina
Status: Completed | Type: Observational
Sponsor: Hospital de Rehabilitacion Manuel Rocca (Other)
Responsible Party: Principal Investigator, Gerardo Candoni, Physical Therapist, Hospital de Rehabilitacion Manuel Rocca
Other Study IDs: 12751
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-06

CONDITIONS: Surveys and Questionnaires; Evaluation of Processes and Results; Healthcare; Evidence-based Clinical Practice; Health Care System; Stroke; Patient Discharge
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: not aplicable — no intervention

SUMMARY:
Introduction Patients who receive care from stroke units are more likely to survive their stroke, become independent, and return home. Decision-making to decide the location of discharge is influenced more by non-clinical factors than clinical ones.

Objective To analyze the factors that are considered for discharge and how stroke patients are measured in stroke units in Argentina by the physicians who make the decisions.

Materials and methods An observational, analytical, cross-sectional survey-type study will be carried out. The recommendations given by the Checklist for Reporting of Survey Studies will be used. It will be intended for all those physicians in Argentina who work in stroke units and discharge.

ELIGIBILITY:
Inclusion Criteria:

* All physicians who in stroke units of Argentina and are in charge of the referral process for hospitalized patients will be included.

Exclusion Criteria:

* All surveys with missing data will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Neurology/Clinical physician/Neurosurgery/Physiatrist/Other
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-03-02 (Actual)

PRIMARY OUTCOMES:
Referral location | 3 months
  It will be qualified as a polytomous qualitative variable (Rehabilitation center/Day hospital/Home/Outpatient clinic/Other)

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica la sagrada familia, Caba, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No